CLINICAL TRIAL: NCT05178615
Title: Investigation of the Effect of Preoperative Education on Postoperative Outcomes in Total Knee Arthroplasty Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Senem Demirdel, Asst Prof, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021-344
Record Dates: First submitted 2021-12-01; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Knee Osteoarthritis; Pain, Postoperative; Kinesiophobia
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative; Kinesiophobia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Experimental): Preoperative education
  Interventions: Other: preoperative education
- control (No Intervention): Traditionally care

INTERVENTIONS:
Other: preoperative education — Education about knee anatomy, patophysiology, total knee arthroplasty surgery, pain neurophysiology, management of pain, the importance of exercise
  Arms: Education group

SUMMARY:
Total knee arthroplasty surgery is a common surgical procedure used in the treatment of patients in the end stages of osteoarthritis. Arthroplasty surgery is a process that creates physical and psychological stress on the patient. Preoperative education can reduce anxiety and improve postoperative outcomes. In the studies on education in the literature, it is seen that there are trainings in the form of seminars, trainings made with video recordings, trainings in the form of brochures. Studies in the literature have shown that training given synchronously (live) by a healthcare professional is more effective in reducing anxiety in one-on-one or small-person groups. Less anxiety does not significantly reduce pain levels, but improves patients' ability to cope with pain and increases their perception of preparedness. Together, these two factors can improve patients' overall experience by increasing their sense of control and comfort.

DETAILED DESCRIPTION:
Studies in the literature define pre-operative education as any educational intervention that aims to improve people's knowledge, health behaviors, and health outcomes before surgery. A 2014 Cochrane© review concluded that pre-operative education provides benefits over standard patient care for hip or knee arthroplasty.

The content of pre-operative education varies, but typical educational materials include information on pre-operative processes, actual steps in the surgical procedure, discharge status, post-operative care, possible surgical and non-surgical complications, answers to frequently asked questions, postoperative pain. The training format consists of one-on-one oral communication, patient group sessions, and a video or booklet. Due to the pandemic process, telerehabilitation methods have become widespread recently. Total knee arthroplasty preoperative trainings conducted to date have been shown to be effective in the form of training given to few people or one-on-one conversations. But to minimize the risk of Covid-19, online education seems to make sense. Researches generally focus on the post-surgical period. However, while the studies emphasized the importance of preoperative education, The investigators did not find any synchronous education in the literature.

Patient satisfaction after joint replacement was found to be directly proportional to meeting expectations for functional outcome and pain. Education given in the preoperative period can affect patient satisfaction by influencing attitudes about patient expectations and pain.

Psychological status has also been reported to be associated with functional outcomes in total knee arthroplasty patients. Fear of movement is an important condition that affects the functionality and recovery of the patient. It has been reported that fear of movement (kinesiophobia) affects early postoperative functional outcomes in total knee arthroplasty patients. Postoperative applications have been shown to be effective on kinesiophobia. However, the investigators could not find any study examining the effect of preoperative education on postoperative outcomes.

The aim of the study is to examine the effect of preoperative education intervention on postoperative pain level, pain beliefs, anxiety and depression, satisfaction, kinesiophobia in total knee arthroplasty patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of noninflammatory arthritis
* Being the first to undergo Total knee arthroplasty surgery,

Exclusion Criteria:

* Lower extremity surgery in the last 1 year,
* Body mass index of 40 and above,
* Revision surgery
* Single compartment replacement
* Psychiatric illness

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain Beliefs Questionnaire | five minutes
  It contains 12 items related to pain beliefs. PBQ-O is an 8-item subscale, and PBQ-P is a 4-item subscale. The organic subscale reflects predominantly organic aspects of pain, with items such as "pain is a result of damage to body tissues" or "experiencing pain is a sign that something is wrong with the body", while the psychological beliefs scale predominantly reflects organic aspects of pain. Reflects the influence of psychological factors on pain, with items such as "worrying makes the pain worse" or "thinking about the pain makes it worse" This assessment will be applied prior to the education given in the pre-operative period. It will be reapplied on the day of discharge in the postoperative period to measure the change after education.
Tampa Scale of Kinesiophoby | Five minutes
  It is a 17-item scale used to measure fear of movement/re-injury. The scale is used to measure injury/re-injury and fear/avoidance parameters in work-related activities. his assessment will be applied prior to the education given in the pre-operative period. It will be reapplied on the day of discharge in the postoperative period to measure the change after education.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | Five minutes
  HAD is a 14-item questionnaire that reliably detects depression and anxiety in a hospital outpatient clinic. his assessment will be applied prior to the education given in the pre-operative period. It will be reapplied on the day of discharge in the postoperative period to measure the change after education.
Numerical Pain Rating Scale | One minute
  Numerical Pain Rating Scale will be used for evaluation of knee pain. On this scale, the severity of pain is graded from 0 to 10. "0" means no pain, "10" means maximum pain. As the score increases, the severity of the pain also increases.This assessment will be applied prior to the education given in the pre-operative period. It will be reapplied on the day of discharge in the postoperative period to measure the change after education.
Patient satisfaction | Six minutes
  Patient satisfaction will be evaluated with expressions created by reviewing the expressions used to evaluate the satisfaction of patients who have previously undergone Total knee arthroplasty.To assess satisfaction, 7 items created by the authors will be scored with a 4-level Likert scale (1=Not at all satisfied, 2=Not satisfied, 3=Satisfied, 4=Very satisfied). The items that evaluate satisfaction are as follows:
  1. "Are you satisfied with your current mobility?"
  2. "Are you satisfied with your current pain situation?"
  3. "Are you satisfied with your current knee movements?"
  4. "Are you satisfied with the current pain level according to your expectations before the operation?"
  5. "Are you satisfied with the information about the post-operative period?"
  6. "Are you satisfied with your sleep quality after the operation?"
  7. "Are you satisfied with the treatment as a whole?"

IPD SHARING:
Plan to Share IPD: No